CLINICAL TRIAL: NCT04270396
Title: Implant Failure and Risk Indicators
Brief Title: Early and Late Implant Failure
Status: Completed | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Joan Takamoli, DDS, Universitat Internacional de Catalunya
Other Study IDs: PER-ECL-2017-04
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Dental Implant Failed; Peri-Implantitis
Keywords: dental implant survival; implant failure; early implant failure; late implant failure
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Presence or absence of implant — We procedure to observed clinically the sample size, to be able to determine if the dental implant was present or no. If the implant was absent we recorded if it was early( prior to restoration) or late ( after prosthesis was delivered).

SUMMARY:
The aim of this study was to evaluate the early and late implant loss rate in a sample of patients who had received implant-supportive restorative therapy in a university setting. Moreover, the study aimed to identify patient- and implant-related variables for implant failure

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old
* Partially or totally edentulous patients with at least one implant placed at the university and at least 7 years before.
* Cemented, screwed, or mechanically retained prosthesis.
* Single and partial prostheses, as well as complete arch prosthesis (fixed and removable).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: A sample of men and women over 18 years old, which they had received an implant-supportive restorative therapy in a university setting throughout a period of at least 7 years.
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Implant survival | October 2017 to March 2019
  Early implant loss and late implant loss

SECONDARY OUTCOMES:
Implant failure | October 2017 to March 2019
  biological and mechanical complications

CONTACTS AND LOCATIONS:
Overall Officials: Joan Takamoli, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Joan, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided